CLINICAL TRIAL: NCT03612856
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy/Potency of a Single Dose of Xisomab 3G3, Administered at the Beginning of a Regular Hemodialysis Procedure, in Patients With End-Stage Renal Disease on Chronic Hemodialysis
Brief Title: Safety and Efficacy Study of AB023 (Xisomab 3G3) in End Stage Renal Disease Patients on Chronic Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aronora, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3G3-18-02
Record Dates: First submitted 2018-07-11; First posted 2018-08-02 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: End Stage Renal Disease; Thrombosis
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AB023 (xisomab 3G3)- Dose 1 (Experimental): Participants will receive a single dose of 0.25 mg/kg xisomab 3G3.
  Interventions: Drug: AB023- Dose 1
- AB023 (xisomab 3G3)- Dose 2 (Experimental): Participants will receive a single dose of 0.5 mg/kg xisomab 3G3.
  Interventions: Drug: AB023-Dose 2
- placebo (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AB023- Dose 1 — Participants will receive a single dose of 0.25 mg/kg AB023.
  Other Names: xisomab 3G3- Dose 1
  Arms: AB023 (xisomab 3G3)- Dose 1
Drug: AB023-Dose 2 — Participants will receive a single dose of 0.5 mg/kg AB023.
  Other Names: xisomab 3G3- Dose 2
  Arms: AB023 (xisomab 3G3)- Dose 2
Drug: placebo — Participants will receive a single dose of placebo.
  Arms: placebo

SUMMARY:
This study evaluates the safety and efficacy of AB023 (xisomab 3G3) in patients with end stage renal disease on chronic hemodialysis. Two dose levels will be evaluated in two cohorts. Within each cohort the patients will be randomized to receive either AB023 (xisomab 3G3) or placebo (at a ratio of 2:1 active: placebo).

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. ESRD maintained on stable outpatient HD regimen, using an established (> 3 months) and normally functioning, regular flow, uninfected first mature AV fistula (or AV graft) and skin consistent with standard chronic HD access injuries, and HD stability defined as Kt/V ≥ 1.2 within 3 months prior to screening at a healthcare center for > 3 months from screening.
2. On HD regimen at least 3 times per week for a minimum of 3 hours per dialysis session, using a complication-free well maintained AV fistula (or AV graft), expected and plan to continue this throughout and for at least 3 months beyond the study.
3. Is capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements and study related procedures.
4. Willing to be confined to the CRU for the duration of the study, able to comply with all study-related requirements, and able to adhere to study restrictions and visit schedules.
5. Male or female, between 18 and 80 years of age (inclusive) at the time of screening.
6. BMI of ≥ 18 at the time of screening.
7. Considered by the PI to be clinically stable with respect to underlying ESRD, based on medical evaluation that includes medical and surgical history, and a complete physical examination including vital signs, ECG, and clinical laboratory test results at screening. Repeat assessments are permitted for any laboratory, ECG, or vital sign parameter required for enrollment.
8. Female patients must be of non-childbearing potential and must have undergone one of the following:

   * sterilization procedures at least 6 months prior to dosing:
   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
9. Male patients must either be sterile (vasectomy with history of a negative sperm count following the procedure); practice total abstinence from sexual intercourse as the preferred lifestyle (periodic abstinence is not acceptable); use a male condom with any sexual activity; or agree to use a birth control method considered to be appropriate by the Investigator (such as one of the methods identified above for female patients) from the time of screening until 90 days after study drug administration. Male patients must agree not to donate sperm for a period of 90 days after study drug administration.

Exclusion Criteria:

Patients must not be enrolled in the study if they meet any of the following criteria:

1. Documented history of acute vasoocclusive thrombotic event (acute coronary syndrome, stroke or transient ischemic attack, venous thromboembolic event), or vascular access fistula or AV graft failure in the past 3 months.
2. With the exception of unfractionated heparin during HD, concomitant or prior use of anticoagulant/antiplatelet agents (e.g., low molecular weight heparins, warfarin, apixaban, bivalirudin, ticagrelor, edoxaban, dabigatran, rivaroxaban, clopidogrel, prasugrel, ticlopidine, eptifibatide, tirofiban, dipyridamole, diclofenac, and all other NSAIDs) that may affect hemostasis for 2 weeks prior to check-in on Day -8 and throughout the study.
3. Use of unfractionated heparin for HD sessions from check-in on Day -8 and throughout the study.
4. Any clinically significant (CS) concomitant disease or condition (including treatment for such conditions) that, in the opinion of the PI, could either interfere with the study drug, compromise interpretation of study data, or pose an unacceptable risk to the patient.
5. Any other CS abnormalities in laboratory test results at screening that would, in the opinion of the PI, increase the patient's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
6. Pregnant (positive pregnancy test) at screening or check-in on Day -8. If serum human chorionic gonadotropin (hCG) pregnancy test results are indeterminate, follow-up testing should be performed to determine eligibility.

   All female patients will not be pregnant and will have a negative pregnancy test at screening and check-in on Day -8, with the following exception: females receiving dialysis with an indeterminate pregnancy test result or persistently low hCG resulting in a false positive pregnancy test may be included in the study at the discretion of the PI. Postmenopausal patients with a result outside the postmenopausal range or an indeterminate pregnancy test will undergo additional testing with FSH to confirm postmenopausal status prior to study enrollment.
7. Treatment with another investigational drug or device study within 30 days (or 5 half lives, whichever is longer) prior to check-in on Day -8.
8. Acute illness that is considered by the PI to be CS within 2 weeks of check-in on Day 8.
9. Currently have established underlying inherited or acquired symptomatic bleeding disorders and/or are at risk for excessive bleeding per PI judgment or current active bleeding (e.g., gastrointestinal, intracranial), aside from minor bleeding from the puncture site on the AV fistula or AV graft, which would be expected to occur during the dialysis procedure, with the following values:

   * Platelet count < 100,000 cells/mm3 (if < 100,000 but > 75,000 cells/mm3, with permission of PI and medical monitor) at screening
   * INR > 1.4 at screening
   * aPTT up to 1.2 x ULN (if >1.2x ULN up to < 1.5 x ULN, with permission of PI and medical monitor) at screening
   * ALT or AST > 2 x ULN at screening
   * Total bilirubin > 1.2 ULN at screening
   * Hemoglobin concentration < 10 g/dL at screening
10. Seated blood pressure < 90/40 mmHg at screening and check-in on Day -8.
11. Exclusion criteria for ECG at screening and check-in on Day -8:

    Heart rate < 45 and > 110 bpm QTcF interval > 500 msec (bpm = beats per minute; msec = milliseconds; QTcF = QT interval corrected using Fridericia's formula)
    * Any significant arrhythmia or conduction abnormality, (including but not specific to atrioventricular block [2nd degree or higher], Wolff Parkinson White syndrome [unless curative radio ablation therapy]), which, in the opinion of the PI and Medical Monitor, could interfere with the safety for the individual patient.
    * Non-sustained or sustained ventricular tachycardia (> 2 consecutive ventricular ectopic beats at a rate of > 1.7/second).
12. History of a CS allergy to recombinant biologic drug, rodents, or a known sensitivity or idiosyncratic reaction to any compound present in xisomab 3G3, its related compounds, or any compound listed as being present in the study formulation.
13. Participate in strenuous exercise from 48 hours prior to check-in on Day -8 and throughout the study.
14. Positive test for drugs of abuse and/or positive alcohol test at screening or check in on Day 8 if not accounted for by a prescription medication. Patients with a positive test based on a prescribed medication may be enrolled.
15. Positive test at screening for hepatitis B surface antigen (HBsAg) or human immunodeficiency virus (HIV). If a patient with ESRD has positive test results for hepatitis C virus (HCV) but liver function tests are otherwise not clinically significant, the patient may be included at the PI's discretion.
16. Receiving blood purification therapy other than HD.
17. Any other reason that would render the patient unsuitable for study enrollment at the discretion of the PI.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All subject-level clinical, laboratory, samples and imaging data as well as protocols, informed consent forms to participate in the trial, data dictionary, and code book will be preserved for data sharing. Shared data will be deidentifed and all raw data generated in connection with this study will be retained by the Investigator's institution.
  All data will be shared with controlled access. Prior to granting access outside of the Sponsor's archive, data will be deidentified by removing all 18 direct identifiers according to HIPAA Privacy Rule's Safe Harbor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data underlying the reported results will be made available 3 months after publication in a peer-reviewed journal for a period of 5 years.
Access Criteria: Potential parties from other organizations can learn about study data and identify whether it could be suitable for their research purposes though summary information (ClinicalTrials.gov, Pubmed) that will be readily available on our website. Requests for data can be made directly to Aronora, Inc.

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Lorentz CU, Tucker EI, Verbout NG, Shatzel JJ, Olson SR, Markway BD, Wallisch M, Ralle M, Hinds MT, McCarty OJT, Gailani D, Weitz JI, Gruber A. The contact activation inhibitor AB023 in heparin-free hemodialysis: results of a randomized phase 2 clinical trial. Blood. 2021 Dec 2;138(22):2173-2184. doi: 10.1182/blood.2021011725. PMID 34086880

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were screened for the study, of which 10 did not meet eligibility criteria. The remaining 27 participants were enrolled. 3 participants terminated the study prior to randomization either by withdrawing consent or at the PI's discretion. The remaining 24 participants were randomized into the study and dosed.
Period: Pre-dose Period
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Started | 8 | 10 | 9
Completed | 8 | 8 | 8
Not Completed | 0 | 2 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Post-dose Period
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (7.59) | 53.1 (5.30) | 52.6 (9.21) | 53.8 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 5
  Male | 7 | 5 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 6 | 21
  White | 0 | 1 | 2 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Treatment-related Adverse Events (TEAEs) and the Number of TEAEs Will be Summarized Using Frequency Counts (Safety and Tolerability)
Description: TEAEs will be determined by physical examination that will include assessment of skin, head, ears, eyes, nose, throat, respiratory system, cardiovascular system, gastrointestinal system, neurological condition, blood and lymphatic systems, and the musculoskeletal system.
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Incidence of Bleeding at the HD Vascular Access Site (Safety and Tolerability)
Description: The number of clinically relevant and non-major bleeding events from the vascular access site. Bleeding from the access site was assessed immediately following decannulation. Pressure was placed on the access site for 10 min. After 10 minutes, the access site was checked for bleeding. If still bleeding, pressure was applied for another 5 minutes and checked again. This was repeated until hemostasis was achieved and the time to hemostasis was recorded. A time greater than 10 min was considered a non-major bleeding event.
Time Frame: Study Days -7, -5, -3 (pre-dose) 1, 3, and 5 (post-dose)
Measure: Number; unit: events
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
events
  Pre-dose hemodialysis days (days -7, -5, -3) | 0 | 5 | 2
  Post-dose hemodialysis days (days 1, 3, 5) | 0 | 5 | 3

3. Primary Outcome: The Number of Subjects With Abnormal Electrocardiogram That is Related to Treatment Will be Summarized Using Frequency Counts (Safety and Tolerability).
Description: 12-lead electrocardiogram measurement. Abnormal electrocardiogram was determined by the study PI. The result was determined to be treatment-related if the abnormal electrocardiogram occurred post-treatment and not pre-treatment. Data from the specified time points (Study Days 6 and 12) were combined by adding the number of participants on each Study Day that showed an abnormal electrocardiogram compared to pre-treatment (Study Day -8 and Study Day 1, pre-dose).
Time Frame: Study Days -8 and 1, pre-dose (pre-treatment) and Study Days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

4. Primary Outcome: The Number of Subjects That Develop Treatment-related Immunogenicity Will be Summarized Using Frequency Counts (Safety and Tolerability).
Description: Immunogenicity measured by the presence of plasma anti-drug antibodies. Plasma anti-drug antibodies were determined by a validated enzyme-linked immunosorbant assay (ELISA) and the titer of anti-drug antibodies present in patient plasma on Study day 12 was compared to the titer of anti-drug antibodies compared to Study day 1, predose.
Time Frame: Study day 1 (predose) and Study Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

5. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Body Temperature, Frequency, and Relation to Treatment Will be Assessed.
Description: Body temperature will be measured in degrees Celsius. Clinically significant changes in body temperature were determined by the study PI. The result was determined to be treatment related if the change in body temperature occurred at any time post-treatment and not pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (1h post-dose), 3, 5, 6, 8, 10, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

6. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Respiratory Rate, Frequency, and Relation to Treatment Will be Assessed.
Description: Respiratory rate will be measured in breaths per minute. Clinically significant changes in respiratory rate were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in respiratory rate occurred post-treatment compared to pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (1h post-dose), 3, 5, 6, 8, 10, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

7. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Blood Pressure (Systolic and Diastolic), Frequency, and Relation to Treatment Will be Assessed.
Description: Systolic and diastolic blood pressure will be measured in mmHg. Clinically significant changes in blood pressure were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in blood pressure occurred post-treatment compared to pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (1h post-dose), 3, 5, 6, 8, 10, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

8. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Heart Rate, Frequency, and Relation to Treatment Will be Assessed.
Description: Heart rate will be measured in beats per minute. Clinically significant changes in heart rate were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in heart rate occurred post-treatment compared to pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (1h post-dose), 3, 5, 6, 8, 10, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

9. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Activated Partial Thromboplastin Time (aPTT), Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Plasma aPTT will be measured in seconds. Clinically significant changes in aPTT were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in aPTT occurred post-treatment compared to pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (3h post-dose), 3, 5, 6, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

10. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Prothrombin Time, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Coagulation Panel.
Description: Prothrombin time will be measured in seconds. Clinically significant changes in prothrombin time were determined by the study PI. The result was determined to be treatment related if the clinically significant changes in prothrombin time occurred post-treatment compared to pre-treatment.
Time Frame: Study days -7, -5, -3, and 1 (pre-treatment) and study days 1 (3h post-dose), 3, 5, 6, and 12 (post-treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

11. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Bilirubin (Total and Direct) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Bilirubin (total and direct) levels in the blood will be measured in mg/dL. Clinically significant changes in bilirubin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in bilirubin occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

12. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alkaline Phosphatase Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Alkaline phosphatase levels in the blood will be measured in U/L. Clinically significant changes in alkaline phosphatase were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in alkaline phosphatase occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

13. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Aspartate Aminotransferase (AST) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: AST levels in the blood will be measured in U/L. Clinically significant changes in aspartate aminotransferase (AST) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in AST occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

14. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Alanine Aminotransferase (ALT) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: ALT levels in the blood will be measured in U/L. Clinically significant changes in alanine aminotransferase (ALT) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in ALT occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

15. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Lactate Dehydrogenase (LDH) Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: LDH levels in the blood will be measured in U/L. Clinically significant changes in lactate dehydrogenase (LDH) were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in LDH occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

16. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Albumin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Albumin levels in the blood will be measured in g/dL. Clinically significant changes in albumin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in albumin occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

17. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Sodium Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Sodium levels will be measured in mEq/L. Clinically significant changes in sodium levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in sodium levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

18. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Potassium Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Potassium levels will be measured in mEq/L. Clinically significant changes in potassium levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in potassium levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

19. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Chloride Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Chloride levels will be measured in mEq/L. Clinically significant changes in chloride levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in chloride levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

20. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Glucose Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Blood glucose levels will be measured in mg/dL. Clinically significant changes in glucose levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in glucose occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

21. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Creatinine Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Serum Chemistry Panel.
Description: Creatinine levels will be measured in mg/dL. Clinically significant changes in creatinine levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in creatinine levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

22. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hemoglobin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hemoglobin levels will be measured in g/dL. Clinically significant changes in hemoglobin were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in hemoglobin occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

23. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Hematocrit Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Hematocrit levels will be measured in %. Clinically significant changes in hematocrit were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in hematocrit occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

24. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Total Leukocyte Counts, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Total leukocyte counts will be measured in 10˄3/uL. Clinically significant changes in total leukocyte count were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in total leukocyte count occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

25. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Differential Leukocyte Counts, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Differential leukocyte counts will be measured in %. Clinically significant changes in differential leukocyte counts were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in differential leukocyte counts occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

26. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Red Blood Cell Count, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Red blood cell count will be measured in 10˄6/uL. Clinically significant changes in red blood cell counts were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in red blood cell counts occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

27. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Platelet Count, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Hematology Panel.
Description: Platelet count will be measured in 10˄3/uL. Clinically significant changes in platelet count were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in platelet count occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

28. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine pH, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: pH of the urine will be measured. Clinically significant changes in urine pH were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine pH occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

29. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Specific Gravity, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Specific gravity of the urine will be evaluated. Clinically significant changes in urine specific gravity were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine specific gravity occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

30. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Protein Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Protein levels in the urine will be evaluated. Clinically significant changes in urine protein levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine protein levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

31. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Glucose Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Glucose levels in the urine will be evaluated. Clinically significant changes in urine glucose levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine glucose levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

32. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Ketone Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Ketone levels in the urine will be evaluated. Clinically significant changes in urine ketone levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine ketone levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

33. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Bilirubin Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Bilirubin levels in the urine will be evaluated. Clinically significant changes in urine bilirubin levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine bilirubin levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

34. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Blood Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Blood levels in the urine will be evaluated. Clinically significant changes in urine blood levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine blood levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

35. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Nitrite Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Nitrite levels in the urine will be evaluated. Clinically significant changes in urine nitrite levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine nitrite levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

36. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Urobilinogen Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Urobilinogen levels in the urine will be evaluated. Clinically significant changes in urine urobilinogen levels were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine urobilinogen levels occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

37. Primary Outcome: The Number of Subjects With Clinically Significant Changes in Urine Leukocyte Esterase Levels, Frequency, and Relation to Treatment Will be Assessed as Part of a Standard Urinalysis Panel (Unless Patient is Anuric).
Description: Leukocyte esterase levels in the urine will be evaluated. Clinically significant changes in urine leukocyte esterase were determined by the study PI. The result was determined to be treatment-related if the clinically significant changes in urine leukocyte esterase occurred post-treatment compared to pre-treatment.
Time Frame: Study day 1 (pre-treatment), and study days 6 and 12 (post-treatment)
Population: Only one subject in the study was able to produce urine. The rest were anuric.
Measure: Count of Participants; unit: Participants
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 0 | 1 | 0
Participants | 0 | 0 | 0

38. Secondary Outcome: Hemodialysis Efficiency as Measured by Frequency of Clotting on the Dialysis Filters and Circuit (Pharmacodynamic Outcome).
Description: Assessment of thrombus accumulation in the dialyzer cartridge measured by visual inspection.
Time Frame: At each hemodialysis session (pre-dose days: study day -7, -5, -3, and post-dose dose days: study day 1, 3, and 5)
Measure: Number; unit: Complete occlusions of filter
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
Complete occlusions of filter
  Pre-dose hemodialysis (days -7, -5, -3) | 2 | 4 | 1
  Post-dose hemodialysis (days 1, 3, 5) | 0 | 0 | 0

39. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Urea Nitrogen (BUN) Levels (Pharmacodynamic Outcome).
Description: Assessment of BUN (mg/dL) before and after hemodialysis as urea reduction ratio (URR), %.
Time Frame: 21 days
Population: In a few instances, the pre- and post-dialysis values appeared to be switched and were excluded from the summary statistics or a value was missing or not reportable.
Measure: Mean (Standard Deviation); unit: URR (%)
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
URR (%)
  Pre-dose Day -7 | 66.53 (4.734) | 70.59 (7.361) | 69.61 (6.452)
  Pre-dose Day -5 | 64.98 (4.927) | 70.36 (5.759) | 70.37 (6.015)
  Pre-dose Day -3: number analyzed (Participants) | 7 | 7 | 8
  Pre-dose Day -3 | 66.67 (6.624) | 67.04 (10.576) | 68.73 (6.378)
  Post-dose Day 1 | 67.82 (6.201) | 69.37 (10.440) | 71.36 (6.098)
  Post-dose Day 3: number analyzed (Participants) | 8 | 7 | 8
  Post-dose Day 3 | 67.47 (5.496) | 72.14 (5.613) | 70.33 (6.877)
  Post-dose Day 5 | 69.63 (5.972) | 71.42 (6.944) | 71.86 (5.864)
  Post-dose Day 12 | 65.66 (8.039) | 72.34 (6.749) | 70.98 (6.315)

40. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Urea Nitrogen (BUN) Levels (Pharmacodynamic Outcome), KtV.
Description: Assessment of BUN (mg/dL) before and after hemodialysis as KtV (mL/min).
Time Frame: 21 days
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mL/min
  Pre-dose Day -7 | 1.312 (0.1537) | 1.449 (0.3051) | 1.413 (0.2359)
  Pre-dose Day -5 | 1.250 (0.1615) | 1.402 (0.2467) | 1.432 (0.2253)
  Pre-dose Day -3: number analyzed (Participants) | 7 | 7 | 8
  Pre-dose Day -3 | 1.330 (0.2078) | 1.337 (0.3887) | 1.347 (0.2239)
  Post-dose Day 1 | 1.386 (0.2311) | 1.438 (0.4005) | 1.492 (0.2424)
  Post-dose Day 3 | 1.399 (0.1894) | 1.509 (0.2505) | 1.431 (0.2482)
  Post-dose Day 5: number analyzed (Participants) | 8 | 7 | 7
  Post-dose Day 5 | 1.393 (0.1841) | 1.494 (0.3209) | 1.451 (0.2383)
  Post-dose Day 12 | 1.253 (0.2267) | 1.527 (0.3107) | 1.478 (0.2480)

41. Secondary Outcome: Hemodialysis Efficiency as Measured by Blood Potassium Levels (Pharmacodynamic Outcome).
Description: Assessment of plasma potassium (mEq/L) before and after hemodialysis. The reduction of plasma potassium (before hemodialysis minus after hemodialysis) is reported in mEq/L).
Time Frame: 21 days
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: mEq/mL
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
mEq/mL
  Pre-dose Day -7 | 1.68 (0.648) | 1.60 (0.595) | 1.69 (0.722)
  Pre-dose Day -5: number analyzed (Participants) | 6 | 8 | 8
  Pre-dose Day -5 | 1.57 (0.769) | 1.44 (0.802) | 1.71 (0.770)
  Pre-dose Day -3: number analyzed (Participants) | 7 | 7 | 8
  Pre-dose Day -3 | 1.44 (0.668) | 1.41 (0.308) | 1.63 (0.590)
  Post-dose Day 1 | 2.11 (0.405) | 1.66 (0.862) | 2.05 (1.207)
  Post-dose Day 3: number analyzed (Participants) | 8 | 7 | 8
  Post-dose Day 3 | 2.11 (0.603) | 1.81 (0.521) | 1.58 (0.861)
  Post-dose Day 5: number analyzed (Participants) | 8 | 7 | 7
  Post-dose Day 5 | 2.00 (0.504) | 1.70 (0.751) | 1.99 (0.734)
  Post-dose Day 12 | 1.24 (0.566) | 1.45 (0.389) | 1.39 (0.813)

42. Secondary Outcome: Hemodialysis Efficiency as Measured by Length of the Hemodialysis Session (Pharmacodynamic Outcome).
Description: The length of each hemodialysis session will be recorded.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
minutes
  Pre-dose Day -7 | 235 (8.44) | 237 (4.84) | 240 (0.00)
  Pre-dose Day -5 | 240 (7.75) | 234 (8.89) | 240 (0.00)
  Pre-dose Day -3 | 242 (4.60) | 239 (3.54) | 240 (0.00)
  Post-dose Day 1 | 233 (15.9) | 232 (15.6) | 240 (0.00)
  Post-dose Day 3 | 240 (0.00) | 235 (12.6) | 240 (0.00)
  Post-dose Day 5 | 240 (0.00) | 239 (1.77) | 240 (0.00)
  Post-dose Day 12 | 232 (14.1) | 239 (3.18) | 240 (0.00)

43. Secondary Outcome: The Effect of a Single Intravenous Dose of Xisomab 3G3 on the Activated Partial Thromboplastin Time (aPTT) (Pharmacodynamic Outcome).
Description: Activated partial thromboplastin time (aPTT) will be measured as a pharmacodynamic marker and the change from baseline will be summarized using descriptive statistics. aPTT is a clotting assay that measures how long it takes for blood to clot after clotting is activated by an intrinsic coagulation pathway activator such as kaolin.
Time Frame: Study day 1 predose and 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48, 96, 120, 168, 216, and 264 hours after dosing
Population: In one instance, the aPTT value was missing or not reportable.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
Number analyzed (Participants) | 8 | 8 | 8
seconds
  0h | 39.1 (7.90) | 42.2 (4.84) | 39.1 (4.29)
  0.167h | 82.2 (19.7) | 92.3 (11.8) | 42.5 (9.00)
  0.5h | 80.6 (18.8) | 91.9 (12.8) | 38.2 (5.16)
  1h | 77.9 (22.3) | 91.4 (12.5) | 38.2 (6.08)
  2h | 83.5 (23.3) | 89.9 (11.4) | 38.5 (5.87)
  3h | 90.9 (21.5) | 93.7 (4.5) | 39.3 (6.54)
  4h | 88.9 (21.5) | 96.0 (11.7) | 41.5 (9.15)
  6h | 87.6 (19.9) | 92.5 (10.1) | 39.4 (6.97)
  8h | 75.8 (19.490) | 83.9 (5.2) | 38.1 (4.40)
  12h | 72.2 (17.7) | 86.1 (8.2) | 41.4 (15.7)
  16h | 68.0 (17.9) | 84.1 (9.10) | 40.7 (5.76)
  24h | 69.8 (21.7) | 89.6 (10.1) | 36.9 (5.56)
  48h | 60.9 (20.9) | 85.3 (7.30) | 37.0 (5.01)
  96h: number analyzed (Participants) | 8 | 7 | 8
  96h | 54.3 (10.8) | 83.5 (27.2) | 40.1 (8.25)
  120h | 55.4 (16.3) | 66.3 (16.9) | 46.1 (9.03)
  168h | 41.0 (5.4) | 59.4 (23.3) | 39.8 (9.03)
  216h | 41.8 (5.5) | 52.6 (17.2) | 39.0 (8.19)
  264h | 44.2 (8.019) | 46.6 (9.94) | 39.6 (5.87)

44. Secondary Outcome: The Maximum Plasma Concentration (Cmax) of Xisomab 3G3 After a Single Injection Will be Measured in Each Patient (Pharmacokinetic Outcome).
Description: Maximum plasma concentration of xisomab 3G3
Time Frame: 14 days
Population: One subject (0.25 mg/kg xisomab 3G3) was excluded from the summary statistics since the 0.17 hr Xisomab 3G3 concentration was suspected to be an outlier.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 7 | 8
ng/mL | 1918 (120.6) | 7557 (33.5)

45. Secondary Outcome: The Time to Reach Maximum Plasma Concentrations of Xisomab 3G3 (Tmax) After a Single Injection Will be Measured in Each Patient (Pharmacokinetic Outcome).
Description: The time to reach maximum plasma concentrations of xisomab 3G3 after a single injection.
Time Frame: 14 days
Population: as for outcome 44
Measure: Median (Full Range); unit: hours
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 7 | 8
hours | 0.167 [0.167 to 3.00] | 0.750 [0.167 to 2.00]

46. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Non-zero Concentration (AUC0-t) After a Single Injection of Xisomab 3G3 Will be Calculated for Each Patient (Pharmacokinetic Outcome)
Description: The area under the plasma concentration-time curve from time 0 to the last measurable non-zero concentration.
Time Frame: 14 days
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 7 | 7
ng*hr/mL | 22330 (214.7) | 256300 (46.9)

47. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) After a Single Injection of Xisomab 3G3 Will be Calculated for Each Patient (Pharmacokinetic Outcome).
Description: The area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) is calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: 14 days
Population: One subject (0.25 mg/kg xisomab 3G3) was excluded from the summary statistics since the 0.17 hr Xisomab 3G3 concentration was suspected to be an outlier. One subject (0.25 mg/kg xisomab 3G3) had an AUC%extrap that was very high (63%) and therefore was excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
ng*hr/mL | 39010 (101.5) | 273200 (54.6)

48. Secondary Outcome: The Percent of AUC0-inf Extrapolated (AUC%Extrap) After a Single Injection of Xisomab 3G3 Will be Calculated for Each Patient (Pharmacokinetic Outcome).
Description: The percent of AUC0-inf extrapolated (AUC%extrap) is calculated by (1-AUC0-t/AUC0-inf)*100. AUC%extrap represents the fraction of the calculated total area under the curve that was extrapolated after the last measured time point.
Time Frame: 14 days
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: percent of AUC that was extrapolated
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
percent of AUC that was extrapolated | 13.55 (11.619) | 5.846 (8.0195)

49. Secondary Outcome: The Apparent First Order Terminal Elimination Rate Constant (Kel) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Subject (Pharmacokinetic Outcome).
Description: The apparent first order terminal elimination rate constant will be calculated from a semi-log plot of the plasma concentration versus time curve. The parameter will be calculated by linear least squares regression analysis using the maximum number of points in the terminal log linear phase (e.g., three or more non zero plasma concentrations).
Time Frame: 14 days
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
1/hr | 0.08800 (0.073260) | 0.03027 (0.010510)

50. Secondary Outcome: The Apparent First Order Terminal Elimination Half-life (T1/2) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Patient (Pharmacokinetic Outcome).
Description: The apparent first order terminal elimination half-life will be calculated as 0.693/Kel.
Time Frame: 14 days
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
hours | 11.125 (5.3961) | 27.082 (15.1722)

51. Secondary Outcome: The Apparent Total Plasma Clearance (CL) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Patient (Pharmacokinetic Outcome).
Description: The apparent total plasma clearance will be calculated as [Dose/AUC0-inf].
Time Frame: 14 days
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
mL/hr | 773.6 (612.47) | 155.0 (42.374)

52. Secondary Outcome: The Total Apparent Volume of Distribution (Vss) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Patient (Pharmacokinetic Outcome).
Description: The total apparent volume of distribution (Vss) will be calculated as the mean residence time x clearance.
Time Frame: 14 days
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2
Number analyzed (Participants) | 6 | 8
mL | 9945 (5014.8) | 5498 (793.78)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study check in (Day -8) through the final follow up (Day 12) for a total of 21 days.
Arm/Group | AB023 (Xisomab 3G3)- Dose 1 | AB023 (Xisomab 3G3)- Dose 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB023 (Xisomab 3G3)- Dose 1 (N=8) | AB023 (Xisomab 3G3)- Dose 2 (N=8) | Placebo (N=8)
Viral gastroenteritis (Infections and infestations) | 2 (2) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Aronora, Inc. shall retain title to and the right to publish all documentation, records, raw data, specimens, or other work product generated in connection with this study. Such publications shall not be made by the PI or Celerion without the prior written consent of Aronora, Inc.

DOCUMENTS (3):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03612856/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03612856/SAP_001.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03612856/ICF_002.pdf